CLINICAL TRIAL: NCT04390113
Title: Phase 3 Multicenter, Double-Blind, Placebo-Controlled Trial of Viralym-M (ALVR105) for the Treatment of Patients With Virus-Associated Hemorrhagic Cystitis After Allogeneic Hematopoietic Cell Transplant (HCT)
Brief Title: Study to Evaluate Viralym-M (ALVR105) for the Treatment of Virus-Associated Hemorrhagic Cystitis (HC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study discontinued as DSMB determined it was futile. No safety concerns were noted.
Sponsor: AlloVir (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVM-003-HC
Record Dates: First submitted 2020-05-12; First posted 2020-05-15 (Actual); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: BK Virus Infection; Hemorrhagic Cystitis
Keywords: Allogeneic Hematopoietic Cell Transplant; ALVR105; Posoleucel
MeSH Terms: conditions — Cystitis, Hemorrhagic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Administered as 2-4 milliliter infusion, visually identical to Posoleucel (ALVR105)
  Interventions: Biological: Placebo
- Posoleucel (ALVR105) (Experimental): Administered as 2-4 milliliter infusion, visually identical to placebo
  Interventions: Biological: Posoleucel (ALVR105)

INTERVENTIONS:
Biological: Posoleucel (ALVR105) — Administered as 2-4 milliliter infusion, visually identical to placebo
  Arms: Posoleucel (ALVR105)
Biological: Placebo — Administered as 2-4 milliliter infusion, visually identical to Posoleucel (ALVR105)
  Arms: Placebo

SUMMARY:
Study to Evaluate Viralym-M (ALVR105) for the Treatment of Virus-Associated Hemorrhagic Cystitis (HC).

DETAILED DESCRIPTION:
The study hypothesis is that the administration of posoleucel (ALVR105) to patients with virus-associated HC will demonstrate superiority for the time to resolution of HC (as measured by resolution of macroscopic hematuria) compared to patients treated with placebo. The primary hypothesis will be tested in patients with BK virus (BKV) viruria to demonstrate superiority over placebo in this population (BK Intent-to-Treat [ITT] Population). A supplementary analysis will be conducted in all patients with any virus-associated HC (cytomegalovirus [CMV], human herpesvirus 6 [HHV-6], Epstein-Barr virus [EBV], JC virus [JCV], and/or adenovirus [AdV]) in order to evaluate efficacy in this broader population (ITT Population).

ELIGIBILITY:
Key Inclusion Criteria

Participants must meet all of the following criteria in order to be eligible to participate in the study:

* Male or female ≥1 year of age.
* Had an allogeneic hematopoietic cell transplant (HCT) performed ≥21 days and ≤1 year prior to randomization.
* Myeloid engraftment confirmed, defined as an absolute neutrophil count ≥500/mm³ for 3 consecutive laboratory values obtained on different days, and platelet count >10,000/mm³ at the time of randomization.
* Diagnosed with HC based on the following criteria (all 3 criteria must be met):

  1. Clinical signs and/or symptoms of cystitis.
  2. Grade ≥3 hematuria, defined as macroscopic hematuria with visible clots.
  3. Viruria with ≥1 target virus (ie, BKV, JCV, AdV, CMV, EBV, and/or HHV-6).
* At least 1 identified, suitably matched posoleucel (ALVR105) cell line for infusion is available.

Key Exclusion Criteria

Participants who meet any of the following criteria will be excluded from participation in the study:

* Ongoing therapy with high-dose systemic corticosteroids (ie, prednisone dose >0.5 mg/kg/day or equivalent).
* Therapy with antithymocyte globulin, alemtuzumab (Campath-1H), or other immunosuppressive T cell-targeted monoclonal antibodies ≤28 days before randomization.
* Evidence of active Grade >2 acute graft versus host disease (GVHD).
* Uncontrolled or progressive bacterial or fungal infections.
* Uncontrolled or progressive viral infections not targeted by posoleucel (ALVR105).
* Uncontrolled or progressive EBV-associated post-transplant lymphoproliferative disorder.
* Known or presumed pneumonia secondary to any organism that is not considered to be well-controlled by antimicrobial therapy.
* Pregnant or lactating or planning to become pregnant.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (56):
- United States (25):
  - City of Hope National Medical Center, Duarte, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Yale University School of Medicine - Yale Cancer Center, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Moffitt, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospital - Kansas City, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University Medical Center (OSUMC), Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- France (5):
  - CHU de Lille - Hopital Claude Huriez, Lille
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - AP-HP Hopital Saint-Louis, Paris
  - HCL Centre Hospitalier Lyon Sud, Pierre-Bénite
  - IUCT-Oncopole, Toulouse
- Italy (7):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria Integrata Verona-Ospedale Borgo Trento, Verona
- South Korea (7):
  - Chonnam National University Hwasun Hospital, Jeongnam
  - Asan Medical Center, Seoul
  - Pusan National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (4):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitari i Politecnic La Fe, Valencia
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (7):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Queen Elizabeth University Hospital - Glasgow, Glasgow
  - Great Ormond Street Hospital for Children, London
  - Hammersmith Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - University College London Hospital, London
  - Nottingham University Hospitals, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tzannou I, Papadopoulou A, Naik S, Leung K, Martinez CA, Ramos CA, Carrum G, Sasa G, Lulla P, Watanabe A, Kuvalekar M, Gee AP, Wu MF, Liu H, Grilley BJ, Krance RA, Gottschalk S, Brenner MK, Rooney CM, Heslop HE, Leen AM, Omer B. Off-the-Shelf Virus-Specific T Cells to Treat BK Virus, Human Herpesvirus 6, Cytomegalovirus, Epstein-Barr Virus, and Adenovirus Infections After Allogeneic Hematopoietic Stem-Cell Transplantation. J Clin Oncol. 2017 Nov 1;35(31):3547-3557. doi: 10.1200/JCO.2017.73.0655. Epub 2017 Aug 7. PMID 28783452
- [Derived] Vasileiou S, Kuvalekar M, Velazquez Y, Watanabe A, Leen AM, Gilmore SA. Phenotypic and functional characterization of posoleucel, a multivirus-specific T cell therapy for the treatment and prevention of viral infections in immunocompromised patients. Cytotherapy. 2024 Aug;26(8):869-877. doi: 10.1016/j.jcyt.2024.03.012. Epub 2024 Mar 19. PMID 38597860

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from March 2021 to Jan 2024 across 57 study centers in the United States, Canada, France, Italy, Spain, Sweden, the United Kingdom and South Korea.
Pre-assignment Details: Overall 144 participants were screened and a total of 97 participants were randomized in the study.
Groups:
- Posoleucel (ALVR105): All participants received 2 infusions of either posoleucel (PSL) or placebo separated by 14 (±3) days. Administering the second infusion as early as 11 days after the first infusion was encouraged if feasible. Participants who weighed <40 kg at the time of screening received 2×10^7 PSL cells (or placebo), while those who weighed ≥40 kg at the time of screening received 4×10^7 PSL cells (or placebo). All infusions were administered intravenously (IV) (via peripheral or central line) over approximately 5 minutes as a slow push.
- Placebo: All participants received 2 infusions of either PSL or placebo separated by 14 (±3) days. Administering the second infusion as early as 11 days after the first infusion was encouraged if feasible. Participants who weighed <40 kg at the time of screening received 2×10^7 PSL cells (or placebo), while those who weighed ≥40 kg at the time of screening received 4×10^7 PSL cells (or placebo). All infusions were administered (IV) (via peripheral or central line) over approximately 5 minutes as a slow push.
Period: Overall Study
Arm/Group | Posoleucel (ALVR105) | Placebo
Started | 57 | 40
Completed | 37 | 26
Not Completed | 20 | 14
Not completed — Not Treated | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Death | 2 | 1
Not completed — Physician Decision | 1 | 3
Not completed — Study Terminated by Sponsor | 5 | 3
Not completed — Withdrawal by Subject | 10 | 5
Not completed — Other | 1 | 0
Not completed — Missing | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Posoleucel (ALVR105); Placebo: All participants received 2 infusions of either PSL or placebo separated by 14 (±3) days. Administering the second infusion as early as 11 days after the first infusion was encouraged if feasible. Participants who weighed <40 kg at the time of screening received 2×10^7 PSL cells (or placebo), while those who weighed ≥40 kg at the time of screening received 4×10^7 PSL cells (or placebo). All infusions were administered (IV) (via peripheral or central line) over approximately 5 minutes as a slow push.
- Total: Total of all reporting groups
Arm/Group | Posoleucel (ALVR105) | Placebo | Total
Number analyzed (Participants) | 57 | 40 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (16.59) | 47.0 (16.60) | 45.8 (16.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 38 | 24 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 7 | 20
  Not Hispanic or Latino | 38 | 30 | 68
  Unknown or Not Reported | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 9 | 2 | 11
  White | 33 | 30 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to Resolution of Macroscopic Hematuria
Description: Time to macroscopic hematuria resolution is calculated from time of randomization to the first date of observed macroscopic hematuria resolution. Kaplan-Meier estimates reported as median number of days to resolution. Participants were censored at the last follow-up time of any participant in the ITT population if they took definitive therapies to stop bladder bleeding or received treatment for hemorrhagic cystitis with non-PSL VSTs before achieving resolution or deceased. Participants were also censored at last follow up if they failed to achieve resolution by end of study.
Time Frame: Up to 24 weeks
Population: BK Intent-to-Treat [ITT] Population: All patients randomized who had BKV in their urine at baseline.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Posoleucel (ALVR105) | Placebo
Number analyzed (Participants) | 48 | 38
Days | 36 [22.0 to 63.0] | 31 [18.0 to 63.0]
Statistical Analysis 1: Comparison: Posoleucel (ALVR105) vs Placebo; Test type: Superiority; p = 0.6253, Log Rank; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.55 to 1.55]

2. Secondary Outcome: Time Until Bladder Pain is Resolved
Time Frame: Until event occurrence through Week 24
Population: Data not collected due to early termination after Data and Safety Monitoring Board (DSMB) futility analysis concluded the study was unlikely to meet its primary endpoint.
Arm/Group | Posoleucel (ALVR105) | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Days in the Hospital for Any Reason
Time Frame: Until event occurrence through Week 24
Population: Data not collected due to early termination after DSMB futility analysis concluded the study was unlikely to meet its primary endpoint.
Arm/Group | Posoleucel (ALVR105) | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Treatment Emergent Acute Graft Versus Host Disease (GVHD)
Description: Grading of acute GVHD is reported according to CTCAE version 5.0 which ranges from Grade 0 (best/no disease) to Grade IV (worst). Participants with Grade I-IV are included.
Time Frame: Up to 24 weeks
Population: Modified ITT Population (mITT): All randomized participants who receive any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105) | Placebo
Number analyzed (Participants) | 57 | 39
Participants | 11 | 9

5. Secondary Outcome: Number of Participants With Treatment Emergent Cytokine Release Syndrome (CRS)
Description: CRS is defined as a supraphysiologic response following any immune therapy that results in the activation or engagement of endogenous or infused T cells and/or other immune effector cells. Symptoms can be progressive, must include fever at the onset, and may include hypotension, capillary leak (hypoxia), and end organ dysfunction.
Time Frame: Up to 24 weeks
Population: mITT: All randomized participants who receive any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105) | Placebo
Number analyzed (Participants) | 57 | 39
Participants | 1 | 0

6. Secondary Outcome: Time to Resolution for All Target Viruses
Time Frame: Until event occurrence through Week 24
Population: as for outcome 3
Arm/Group | Posoleucel (ALVR105) | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Average Daily Bladder Pain
Time Frame: Until event occurrence through Week 6
Population: as for outcome 3
Arm/Group | Placebo | Posoleucel (ALVR105)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: All-cause Mortality was collected for all participants enrolled. Serious and Other (not including serious) Adverse Events were collected for participants who received at least one dose of investigational product.
Arm/Group | Posoleucel (ALVR105) | Placebo
All-Cause Mortality (participants affected / at risk) | 2/57 | 1/40
Serious Adverse Events (participants affected / at risk) | 28/57 | 19/39
Other Adverse Events (participants affected / at risk) | 54/57 | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posoleucel (ALVR105) (N=57) | Placebo (N=39)
Pneumonia (Infections and infestations) | 4 | 1
Viral haemorrhagic cystitis (Infections and infestations) | 2 | 2
COVID-19 pneumonia (Infections and infestations) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 2 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Human herpesvirus 6 encephalitis (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Post-acute COVID-19 syndrome (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 2 | 0
Anuria (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Viral haemorrhagic cystitis (Renal and urinary disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Abdominal pain (General disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 3
Asthenia (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute graft versus host disease in intestine (Immune system disorders) | 2 | 1
Acute graft versus host disease in liver (Immune system disorders) | 0 | 1
Chronic graft versus host disease in intestine (Immune system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Shock haemorrhagic (Vascular disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Lipase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Arterial revascularisation (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Posoleucel (ALVR105) (N=57) | Placebo (N=39)
Pneumonia (Infections and infestations) | 6 | 4
COVID-19 (Infections and infestations) | 6 | 3
Urinary tract infection (Infections and infestations) | 3 | 5
Cytomegalovirus infection reactivation (Infections and infestations) | 3 | 3
Oral candidiasis (Infections and infestations) | 3 | 3
Epstein-Barr virus infection reactivation (Infections and infestations) | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Viral haemorrhagic cystitis (Infections and infestations) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 13 | 8
Nausea (Gastrointestinal disorders) | 11 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 7
Vomiting (Gastrointestinal disorders) | 7 | 2
Constipation (Gastrointestinal disorders) | 3 | 3
Dry mouth (Gastrointestinal disorders) | 4 | 1
Blood creatinine increased (Investigations) | 6 | 6
Neutrophil count decreased (Investigations) | 6 | 5
Platelet count decreased (Investigations) | 7 | 3
White blood cell count decreased (Investigations) | 5 | 3
Aspartate aminotransferase increased (Investigations) | 3 | 3
Blood alkaline phosphatase increased (Investigations) | 2 | 4
Alanine aminotransferase increased (Investigations) | 2 | 3
Blood lactate dehydrogenase increased (Investigations) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 8
Decreased appetite (Metabolism and nutrition disorders) | 6 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 3
Acute graft versus host disease in intestine (Immune system disorders) | 8 | 3
Acute graft versus host disease in skin (Immune system disorders) | 6 | 5
Chronic graft versus host disease in skin (Immune system disorders) | 3 | 3
Chronic graft versus host disease in intestine (Immune system disorders) | 3 | 2
Chronic graft versus host disease in eye (Immune system disorders) | 3 | 1
Pyrexia (General disorders) | 11 | 8
Oedema peripheral (General disorders) | 3 | 4
Fatigue (General disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dysuria (Renal and urinary disorders) | 6 | 2
Acute kidney injury (Renal and urinary disorders) | 3 | 3
Anaemia (Blood and lymphatic system disorders) | 4 | 9
Neutropenia (Blood and lymphatic system disorders) | 6 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3
Hypotension (Vascular disorders) | 6 | 4
Hypertension (Vascular disorders) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Headache (Nervous system disorders) | 2 | 3
Confusional state (Psychiatric disorders) | 3 | 2
Depression (Psychiatric disorders) | 3 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 1
Tachycardia (Cardiac disorders) | 3 | 1
Dry eye (Eye disorders) | 3 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Pericardial effusion (Cardiac disorders) | 3 | 0
Acute graft versus host disease in liver (Immune system disorders) | 1 | 2
Chronic graft versus host disease oral (Immune system disorders) | 3 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 2
Adenovirus infection (Infections and infestations) | 3 | 1
Parainfluenzae virus infection (Infections and infestations) | 2 | 2
Urinary tract infection bacterial (Infections and infestations) | 2 | 2
Cytomegalovirus viraemia (Infections and infestations) | 3 | 0
Blood bilirubin increased (Injury, poisoning and procedural complications) | 1 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 3
C-reactive protein increased (Investigations) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 3
Hallucination (Psychiatric disorders) | 1 | 2
Insomnia (Psychiatric disorders) | 3 | 0
Agitation (Psychiatric disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Haematuria (Renal and urinary disorders) | 4 | 0
Urinary retention (Renal and urinary disorders) | 4 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
AlloVir decided to discontinue the trial on 22-Dec-2023 following a pre-planned DSMB futility analysis concluding the study was unlikely to meet its primary endpoint; no safety concerns were identified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT04390113/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/13/NCT04390113/SAP_001.pdf